CLINICAL TRIAL: NCT02666482
Title: Using Technology to Help Low-income and Latino Smokers Quit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i4Health (Other)
Collaborators: Center for Behavioral Intervention Technologies (Unknown); San Francisco Health Network (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24RT-0027
Record Dates: First submitted 2016-01-21; First posted 2016-01-28 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Smoking Cessation
Keywords: smoking; stop smoking; tobacco use cessation
MeSH Terms: conditions — Smoking Cessation; Smoking; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stop Smoking SF Web App - baseline (Experimental): Online Study 1 will test the data gathering aspects of the proposed web app using a baseline, "usual care" intervention consisting of a static smoking cessation guide, the Guía para Dejar de Fumar, tested in printed form in the Muñoz et al. (1997) study. The print version of the guide yielded an 11% quit rate at 3 months. The investigators will utilize the content of the guide as the main element of the baseline app, so it will serve to estimate baseline utilization and quit rates when this already tested intervention is provided in a web app format. Participants can join the study online by going to: https://stopsmokingsf.org
  Interventions: Behavioral: Stop Smoking SF Web App - baseline

INTERVENTIONS:
Behavioral: Stop Smoking SF Web App - baseline — Smoking cessation web app in Spanish and English. Accessible online at no charge.

SUMMARY:
The Institute for International Internet Interventions for Health (i4Health) at Palo Alto University proposes to develop digital tools specifically designed to help low income English-speaking and Spanish-speaking smokers to quit. The investigators aim to test whether a mobile-based digital intervention designed with systematic input from low-income English- and Spanish-speaking smokers from a public sector health care system can significantly improve its acceptability, utilization, and effectiveness. Using human-centered development methods, the project will involve low-income patients of the San Francisco Health Network in the design of a web app/text messaging tool. The investigators will also use participants input to improve the recruitment and dissemination strategies. i4Health will join forces with the Center for Behavioral Intervention Technologies (CBITs) at Northwestern University to iteratively develop successive versions of the digital interventions informed by our human-centered approach.

The full study involves 4 successive outcome studies testing the effectiveness of the Stop Smoking San Francisco web app.

The first three are single-group non-randomized pre-post studies with 1, 2, and 3-month follow-ups. These will test gradually improved versions of the app.

The fourth study will involve a randomized trial comparing the initial version (the baseline version) of the web app to the final version of the web app, to determine if the final version is significantly better than the baseline version in terms of increased utilization and abstinence rates.

To join this study, go to: https://stopsmokingsf.org

DETAILED DESCRIPTION:
The project involves three specific aims:

Specific Aim #1: Human-centered development of an English/Spanish smoking cessation web app. The investigators will develop iterative versions of a digital smoking cessation tool (a web app with text messaging components) that is highly responsive to the needs and preferences of low-income English- and Spanish-speaking smokers. Development will take place with systematic input from patients who are part of the San Francisco Health Network (SFHN). The SFHN serves 70,000 members, most of whom are low-income individuals.

Specific Aim #2: Improvement of dissemination strategies. Input from SFHN patients will identify effective ways of reaching and encouraging low-income English- and Spanish-speaking smokers to use the digital smoking cessation interventions to be developed. This information will support ongoing dissemination and implementation efforts beyond the grant period.

Specific Aim #3: Evaluation of resulting smoking cessation web app. Researchers will evaluate the effectiveness of the successive versions of the resulting stop smoking web app by recruiting smokers at two levels: a) within the SFHN, and b) throughout the state of California, culminating with an online randomized controlled trial. Increased effectiveness will be defined as 1) increased utilization of the web app and 2) higher abstinence rates than those obtained by a baseline "usual care" web app.

ELIGIBILITY:
Inclusion Criteria:

* English speaking (ES) and Spanish speaking (SS)

Exclusion Criteria:

* Not a smoker

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1107 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
7-day Quit rate | 1 Month

SECONDARY OUTCOMES:
Utilization of web app: Number of times web app screens are accessed and data entered | 1 month
  Number of times web app screens are accessed and data entered

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F. Munoz, Ph.D., Principal Investigator — Director, i4Health, Palo Alto University
Locations (1):
- Palo Alto University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Munoz RF, Marin BV, Posner SF, Perez-Stable EJ. Mood management mail intervention increases abstinence rates for Spanish-speaking Latino smokers. Am J Community Psychol. 1997 Jun;25(3):325-43. doi: 10.1023/a:1024676626955. PMID 9332966
- [Background] Muñoz, R. F., Bunge, E. L., Chen, K., Schueller, S. M., Bravin, J. I., Shaughnessy, E. A., & Pérez-Stable, E. J. (2015). Massive Open Online Interventions: A novel model for delivering behavioral-health services worldwide. Clinical Psychological Science. Advance online publication. doi: 10.1177/2167702615583840
- [Derived] Munoz RF, Bunge EL, Barrera AZ, Wickham RE, Lee J. Using Behavioral Intervention Technologies to Help Low-Income and Latino Smokers Quit: Protocol of a Randomized Controlled Trial. JMIR Res Protoc. 2016 Jun 14;5(2):e127. doi: 10.2196/resprot.5355. PMID 27302623